CLINICAL TRIAL: NCT06136871
Title: Cognitive Strategy Training in Post-COVID-19 Syndrome: A Feasibility Trial
Brief Title: Cognitive Rehabilitation in Post-COVID-19 Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Anna Boone, Assistant Professor, Occupational Therapy, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2096158; R21HD112373-01 (NIH)
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Post-COVID-19 Syndrome
Keywords: covid-19; metacognition; cognition; telehealth; activities of daily living
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: After baseline assessment, subjects will be randomized to one of two groups: (1) a 10-session Cognitive Orientation to daily Occupational Performance (CO-OP) intervention; or (2) a 10-session inactive control group.
Who Masked: Outcomes Assessor
Masking Description: All outcomes assessors will be blinded to participant study group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Orientation to daily Occupational Performance (CO-OP) (Experimental): Each CO-OP session will last 45 minutes and subjects will complete one session per week over the course of 10 weeks. All sessions will be delivered remotely via the Zoom platform.
  Interventions: Behavioral: CO-OP Procedures
- Inactive Control Group (Other): Subjects will complete one session per week over the course of 10 weeks. All sessions will be delivered remotely via the Zoom platform.
  Interventions: Behavioral: Inactive Control Group

INTERVENTIONS:
Behavioral: CO-OP Procedures — CO-OP is a metacognitive strategy training intervention that will be used in this study. First, five functional, everyday life goals are identified collaboratively by the participant and interventionist. In the second meeting, we introduce the approach to the subject and teach the global cognitive strategy (i.e., GOAL-PLAN-DO-CHECK). In all subsequent sessions, this strategy is used as the main problem-solving framework to facilitate skill acquisition.The subject identifies a GOAL, and then is guided by the therapist to discover a PLAN to potentially achieve the goal. The subject is then asked to DO the plan (if feasible during the therapy session otherwise asked to complete at home prior to the next treatment session), and subsequently to CHECK to see if the plan worked, i.e. the goal was achieved. This process is repeated until satisfactory performance is met for each established goal.
  Arms: Cognitive Orientation to daily Occupational Performance (CO-OP)
Behavioral: Inactive Control Group — An inactive control group will be used to control for maturation and testing effects. Weekly contact will be made via teleconferencing to (1) maintain study engagement, (2) introduce weekly social contact with researchers, mimicking some of the potential incidental effects of the experimental group, and (3) ascertain what, if any, additional steps participants have taken to reduce PCS symptoms. The content of each of these meetings will be tracked in intervention notes. Each contact will be recorded for fidelity monitoring to ensure all active ingredients of the CO-OP intervention are avoided.
  Arms: Inactive Control Group

SUMMARY:
The first aim of this study is to determine the feasibility of delivering CO-OP remotely to individuals experiencing cognitive impairments that limit everyday activities in post-COVID-19 syndrome (PCS). The second aim of this study is to assess the effect of CO-OP on activity performance, subjective and objective cognition, and quality of life in a sample of individuals with PCS. The research team hypothesizes that effect size estimations will indicate that CO-OP will have a greater positive effect, compared to an inactive control group, on activity performance, subjective and objective cognition, and quality of life in a sample of individuals who self-report PCS and cognitive impairment.

DETAILED DESCRIPTION:
Post-COVID-19 symptoms (PCS) cognitive symptoms require the rehabilitation community to investigate ways to: (1) reduce the functional impact of the symptoms on daily life and (2) support individuals with PCS to establish new habits to improve and maintain health. While the cognitive impairment associated with PCS has not been well evaluated, it is similar of cognitive symptoms seen in other conditions. Metacognitive strategy training (MCST) approaches are an evidence-based practice standard for improving capacity to self-manage chronic cognitive symptoms and reduce their functional impact on everyday life activities.

The CO-OP approach is an MCST intervention in which participants are taught a general cognitive strategy that can be applied in known and novel contexts to devise task specific strategies for engaging in an activity. Existing evidence with other populations suggests that CO-OP has more of a positive effect on improving activity performance and cognition than remediation/retraining-based approaches. These effects have been demonstrated in individuals with mild cognitive impairment that mirrors that found in PCS. The overall research hypothesis is that CO-OP can feasibly be administered remotely and will improve activity performance, subjective and objective cognitive function, and quality of life in individuals with PCS.

ELIGIBILITY:
Inclusion Criteria:

* self-reported cognitive symptoms persisting for at least 6 weeks following COVID-19 infection (Cognitive Failures Questionnaire (CFQ) score >43)
* self-identified activity performance goals per the Canadian Occupational Performance Measure (COPM)
* documented prior diagnosis of COVID-19
* read, write, and speak English fluently
* ability to provide valid informed electronic consent

Exclusion Criteria:

* diagnosis of severe neurological or psychiatric condition(s)
* dementia symptoms as indicated by a score of <23 on the Montreal Cognitive Assessment (MoCA)
* untreated sleep apnea (≥5 on the STOPBANG)
* prior cancer treatment
* severe depressive symptoms (>21 on the Patient Health Questionnaire-9)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | After study completion, an average of 12 weeks
  Number of participants enrolled divided by number of individuals screened
Telehealth Usability Questionnaire (TUQ) | After study completion, an average of 12 weeks
  Measure of telehealth usability from participant's perspective. Self-report Likert scale of 1 (disagree) to 7 (agree)
Acceptability of Intervention Measure (AIM) | After study completion, an average of 12 weeks
  Measure of intervention acceptability. Self-report Likert scale of 1 (completely disagree) to 5 (completely agree)
Intervention Appropriateness Measure (IAM) | After study completion, an average of 12 weeks
  Measure of intervention appropriateness. Self-report Likert scale of 1 (completely disagree) to 5 (completely agree)
Feasibility of Intervention Measure (FIM) | After study completion, an average of 12 weeks
  Measure of intervention feasibility. Self-report Likert scale of 1 (completely disagree) to 5 (completely agree)
Canadian Occupational Performance Measure (COPM) | Pre-intervention (week 0), week 2, week 4, week 6, week 8, and post-intervention (week 12)
  Self-report measure of activity performance. Minimum = 1, Maximum = 10. Higher scores mean better performance.
Retention rate | After study completion, an average of 12 weeks
  Number of participants completing all study procedures divided by number of participants enrolled

SECONDARY OUTCOMES:
Delis-Kaplan Executive Function System (DKEFS)- Color-Word Interference | Pre-intervention (week 0) and post-intervention (week 12)
  Objective measure of inhibition and cognitive flexibility. Consists of 4 conditions (color naming, word reading, inhibition, and inhibition/switching). Therapist records client-corrected errors, noncorrected errors, and total time required for each domain. Increased errors and time indicate potential challenges with inhibition and cognitive flexibility.
Patient-Reported Outcomes Measurement Information System (PROMIS) Cognitive Function | Pre-intervention (week 0) and post-intervention (week 12)
  Self-report measure of cognition. Maximum=5, minimum=1. Higher scores indicate fewer perceived cognitive deficits.
World Health Organization Quality of Life Assessment Instrument (WHOQOL-100) | Pre-intervention (week 0) and post-intervention (week 12)
  Self-report measure of quality of life. Maximum=5, minimum=1. Higher scores indicate greater perceived quality of life.
Cambridge Neuropsychological Test Automated Battery (CANTAB) Rapid Visual Information Processing Subtest | Pre-intervention (week 0) and post-intervention (week 12)
  Objective measure of sustained attention. Other outcomes include latency (speed of response), probability of false alarms, and sensitivity.
CANTAB Spatial Working Memory Subtest | Pre-intervention (week 0) and post-intervention (week 12)
  Objective measure of working memory and strategy.
CANTAB Stockings of Cambridge Subtest | Pre-intervention (week 0) and post-intervention (week 12)
  Objective measure of planning and executive function. Other outcomes include problem-solving ability and time required to complete task.
CANTAB Delayed Matching to Sample Subtest | Pre-intervention (week 0) and post-intervention (week 12)
  Objective measure of short-term visual recognition memory and attention. Other outcomes include latency (speed of response), the number of correct patterns selected and a statistical measure giving the probability of an error after a correct or incorrect response.
CANTAB Paired Associates Learning Subtest | Pre-intervention (week 0) and post-intervention (week 12)
  Objective measure of visual episodic memory. Other outcomes include the errors made by the participant, the number of trials required to locate the pattern(s) correctly, memory scores and stages completed.

CONTACTS AND LOCATIONS:
Overall Officials: Anna E Boone, PhD, OTR/L, Principal Investigator — University of Missouri Occupational Therapy
Locations (1):
- University of Missouri Department of Occupational Therapy, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McEwen S, Polatajko H, Baum C, Rios J, Cirone D, Doherty M, Wolf T. Combined Cognitive-Strategy and Task-Specific Training Improve Transfer to Untrained Activities in Subacute Stroke: An Exploratory Randomized Controlled Trial. Neurorehabil Neural Repair. 2015 Jul;29(6):526-36. doi: 10.1177/1545968314558602. Epub 2014 Nov 21. PMID 25416738
- [Background] Geusgens CA, van Heugten CM, Cooijmans JP, Jolles J, van den Heuvel WJ. Transfer effects of a cognitive strategy training for stroke patients with apraxia. J Clin Exp Neuropsychol. 2007 Nov;29(8):831-41. doi: 10.1080/13803390601125971. PMID 18030634
- [Background] Haskins EC, Cicerone KD, Trexler LE. Cognitive rehabilitation manual: Translating evidence-based recommendations into practice. ACRM Publishing; 2012.
- [Background] Cicerone KD, Dahlberg C, Malec JF, Langenbahn DM, Felicetti T, Kneipp S, Ellmo W, Kalmar K, Giacino JT, Harley JP, Laatsch L, Morse PA, Catanese J. Evidence-based cognitive rehabilitation: updated review of the literature from 1998 through 2002. Arch Phys Med Rehabil. 2005 Aug;86(8):1681-92. doi: 10.1016/j.apmr.2005.03.024. PMID 16084827
- [Background] Dawson DR, Anderson ND, Burgess P, Cooper E, Krpan KM, Stuss DT. Further development of the Multiple Errands Test: standardized scoring, reliability, and ecological validity for the Baycrest version. Arch Phys Med Rehabil. 2009 Nov;90(11 Suppl):S41-51. doi: 10.1016/j.apmr.2009.07.012. PMID 19892074
- [Background] Wolf TJ, Polatajko H, Baum C, Rios J, Cirone D, Doherty M, McEwen S. Combined Cognitive-Strategy and Task-Specific Training Affects Cognition and Upper-Extremity Function in Subacute Stroke: An Exploratory Randomized Controlled Trial. Am J Occup Ther. 2016 Mar-Apr;70(2):7002290010p1-7002290010p10. doi: 10.5014/ajot.2016.017293. PMID 26943113

DOCUMENTS (1):
  • Informed Consent Form: Informed Consent Form Only (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/71/NCT06136871/ICF_000.pdf